CLINICAL TRIAL: NCT05664711
Title: Effect of Stellate Ganglion Block on ME/CFS Symptoms and Metabolites
Brief Title: Effect of Stellate Ganglion Block on ME/CFS
Acronym: SGB_ME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuroversion, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20193104
Record Dates: First submitted 2022-12-12; First posted 2022-12-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Encephalomyelitis, Myalgic; Chronic Fatigue Syndrome; Chronic Fatigue Disorder; Chronic Fatigue and Immune Dysfunction Syndrome; Myalgic Encephalomyelitis; Postviral Fatigue Syndrome; Systemic Exertion Intolerance Disease; Infectious Mononucleosis-Like Syndrome, Chronic; Chronic Fatigue-Fibromyalgia Syndrome
Keywords: ME/CFS; myalgic encephalomyelitis; chronic fatigue syndrome; stellate ganglion block; SGB; cervical sympathetic block; post-exertional malaise; PEM; exertional intolerance; brain fog; orthostatic intolerance
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Mental Fatigue; Orthostatic Intolerance | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Stellate Ganglion Block (Experimental): The stellate ganglion and nearby cervical sympathetic ganglia will be blocked with 10 mL 0.5 percent bupivacaine under ultrasound guidance.
  Interventions: Drug: Bupivacaine Injection

INTERVENTIONS:
Drug: Bupivacaine Injection — Reciprocal unilateral stellate ganglion blocks, separated by at least 16 hours, will be given once per week for three weeks (for a total of 6 blocks).
  This study is not intended to be reported to FDA as a well-controlled study in support of a new indication for bupivacaine or to support any other significant change in the labeling for the drug.
  Other Names: stellate ganglion block

SUMMARY:
The goal of this clinical trial is to study the effects of stellate ganglion block (SGB) in participants with myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). The main questions it aims to answer are:

Does SGB treatment improve symptoms of ME/CFS (e.g. brain fog, fatigue)? Do changes in symptoms go along with changes in blood or saliva?

Participants will receive a total of six blocks over three weeks (one block on each side, one day apart, per week). Prior to treatment and at two points following treatment, participants will complete surveys, take a cognitive (puzzle type) test, and provide blood and saliva for analysis. Participants will measure their heart rate daily using a free smart phone app.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-50 years)
* Female
* ME/CFS (CCC and IOM criteria) duration less than 4 years at time of study enrollment
* Confirmed or suspected viral disease prior to ME/CFS onset (e.g., SARS-CoV-2, Epstein-Barr, Influenza)
* BMI =18-29 kg/m^2
* Ability to read, write and speak English language

Exclusion Criteria:

* Prior SGB treatment
* Allergy to amide local anesthetics (e.g. ropivacaine, bupivacaine)
* Current anticoagulant use
* History of bleeding disorder
* History of glaucoma
* Infection or mass at injection site
* Anatomical abnormalities in C3-T1 region
* Current pregnancy
* Hypertension
* Diabetes (any type)
* Thyroid disease
* History of neck or throat surgeries
* Vocal cord problems or paralysis
* Causalgia/Chronic Regional Pain Syndrome (CRPS)
* Current cancer diagnosis
* Diagnosis of Guillain-Barré syndrome
* Diagnosis of current moderate or severe substance use disorder
* History of neurological disease, seizure, or significant head trauma
* Conditions or disorders (other than ME/CFS) that affect cognitive functioning including stroke, past or present diagnosis of psychosis or psychotic symptoms, diagnosis of bipolar I disorder, or severe depression

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Rating of Symptoms at 2 Weeks | 2 weeks
  The primary objective of the clinical trial is to evaluate whether stellate ganglion block treatment improves the subjective rating of symptoms (severity and frequency) and the amount of limitations to activities. We will measure the change from baseline scores at two weeks for the DePaul Symptom Questionnaire to measure the frequency and severity of symptoms (on a scale of 0 to 4 in which a higher score indicates more frequent or more severe) and the Rand Short Form-36-Physical Fatigue subscale (SF-36PF) to measure the amount of limitations due to symptoms (on a scale of 1-3 in which a higher score indicates less limitation).
Change in Subjective Rating of Symptoms at 2 Months | 2 months
  The primary objective of the clinical trial is to evaluate whether stellate ganglion block treatment improves the subjective rating of symptoms (severity and frequency) and the amount of limitations to activities. We will measure the change from baseline scores at two months for the DePaul Symptom Questionnaire to measure the frequency and severity of symptoms (on a scale of 0 to 4 in which a higher score indicates more frequent or more severe) and the Rand Short Form-36-Physical Fatigue subscale (SF-36PF) to measure the amount of limitations due to symptoms (on a scale of 1-3 in which a higher score indicates less limitation).
Change in Cognitive Function at 2 Weeks | 2 weeks
  The primary objective of the clinical trial is to evaluate whether stellate ganglion block treatment reduces "brain fog" as measured by computerized neurocognitive tests for attention, executive function, and memory. Scores are standardized and scaled to adjust for age and the device on which tests are taken. Scores range from 0 to 200, in which the average score (corresponding to the 50th percentile) is set to 100, and higher scores indicate better cognitive function. Scores are obtained for attention, executive function, and memory. Scores at baseline will be compared to scores at two weeks post-treatment.
Change in Cognitive Function at 2 Months | 2 months
  The primary objective of the clinical trial is to evaluate whether stellate ganglion block treatment reduces "brain fog" as measured by computerized neurocognitive tests for attention, executive function, and memory. Scores are standardized and scaled to adjust for age and the device on which tests are taken. Scores range from 0 to 200, in which the average score (corresponding to the 50th percentile) is set to 100, and higher scores indicate better cognitive function. Scores are obtained for attention, executive function, and memory. Scores at baseline will be compared to scores at two months post-treatment.

SECONDARY OUTCOMES:
Change in Orthostatic Tolerance at 2 Weeks | 2 weeks
  The 10-minute National Aeronautics and Space Administration (NASA) lean test will be used to measure hemodynamic changes during orthostatic challenge (lying down vs. standing up). The study will measure change from baseline at 2 weeks post-treatment.
Change in Orthostatic Tolerance at 2 Months | 2 months
  The 10-minute National Aeronautics and Space Administration (NASA) lean test will be used to measure hemodynamic changes during orthostatic challenge (lying down vs. standing up). The study will measure change from baseline at 2 months post-treatment.
Change in Autonomic Tone at 2 Weeks | 2 weeks
  A wearable device (a ring worn on a finger at night) will be used to measure resting heart rate (beats per minute), heart rate variability (milliseconds), and blood oxygenation (percentage oxygen aka SpO2) during the night and for 5 minutes upon awakening, in combination with a smart phone app, at baseline and two weeks after treatment. These parameters reflect the balance between sympathetic and parasympathetic nervous systems (aka "autonomic tone"). ME/CFS patients are known to have excessive sympathetic tone. Within normal levels, better outcomes are indicated by lower resting heart rate, increased heart rate variability, and increased blood oxygenation.
Change in Autonomic Tone at 2 Months | 2 months
  A wearable device (a ring worn on a finger at night) will be used to measure resting heart rate (beats per minute), heart rate variability (milliseconds), and blood oxygenation (percentage oxygen aka SpO2) during the night and for 5 minutes upon awakening, in combination with a smart phone app, at baseline and two months after treatment. These parameters reflect the balance between sympathetic and parasympathetic nervous systems (aka "autonomic tone"). ME/CFS patients are known to have excessive sympathetic tone. Within normal levels, better outcomes are indicated by lower resting heart rate, increased heart rate variability, and increased blood oxygenation compared to baseline.

OTHER OUTCOMES:
Change in Salivary Cortisol upon Awakening at 2 Weeks | 2 weeks
  Concentration of free cortisol in saliva upon awakening will be measured in micrograms per deciliter (ug/dL) using Enzyme-Linked Immunosorbent Assay (ELISA), at baseline and two weeks after treatment. ME/CFS patients have abnormally low levels of cortisol in general and upon awakening. An increased concentration within the normal range (from 0.007 ug/dL to 0.115 ug/dL) indicates a better outcome.
Change in Salivary Cortisol Upon Awakening at 2 Months | 2 months
  Concentration of free cortisol in saliva upon awakening will be measured in micrograms per deciliter (ug/dL) using Enzyme-Linked Immunosorbent Assay (ELISA), at baseline and two months after treatment. ME/CFS patients have abnormally low levels of cortisol in general and upon awakening. An increased concentration within the normal range (from 0.007 ug/dL to 0.115 ug/dL) indicates a better outcome.
Change in Metabolites at 2 Weeks | 2 weeks
  Plasma will be analyzed by liquid chromatography/mass spectrometry (LC/MS) to determine the levels of 433 hydrophilic metabolites (relative to an unchanging molecule in plasma) at baseline and at two weeks after treatment. ME/CFS patients are known to have abnormally high or low amounts of many metabolites, indicating mitochondrial dysfunction. Changes in abnormal metabolites toward normal values would indicate a better outcome.
Change in Metabolites at 2 Months | 2 months
  Plasma will be analyzed by liquid chromatography/mass spectrometry (LC/MS) to determine the levels of 433 hydrophilic metabolites (relative to an unchanging molecule in plasma) at baseline and at two months after treatment. ME/CFS patients are known to have abnormally high or low amounts of many metabolites, indicating mitochondrial dysfunction. Changes in abnormal metabolites toward normal values would indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L Duricka, PhD, Principal Investigator — Neuroversion, Inc.
Locations (1):
- Neuroversion, Anchorage, Alaska, United States

REFERENCES:
- [Background] Liu LD, Duricka DL. Stellate ganglion block reduces symptoms of Long COVID: A case series. J Neuroimmunol. 2022 Jan 15;362:577784. doi: 10.1016/j.jneuroim.2021.577784. Epub 2021 Dec 8. PMID 34922127
- [Background] van Campen CLMC, Rowe PC, Visser FC. Cerebral blood flow remains reduced after tilt testing in myalgic encephalomyelitis/chronic fatigue syndrome patients. Clin Neurophysiol Pract. 2021 Sep 23;6:245-255. doi: 10.1016/j.cnp.2021.09.001. eCollection 2021. PMID 34667909
- [Background] Campen CLMCV, Rowe PC, Visser FC. Orthostatic Symptoms and Reductions in Cerebral Blood Flow in Long-Haul COVID-19 Patients: Similarities with Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Medicina (Kaunas). 2021 Dec 24;58(1):28. doi: 10.3390/medicina58010028. PMID 35056336
- [Background] Tokumasu K, Honda H, Sunada N, Sakurada Y, Matsuda Y, Yamamoto K, Nakano Y, Hasegawa T, Yamamoto Y, Otsuka Y, Hagiya H, Kataoka H, Ueda K, Otsuka F. Clinical Characteristics of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) Diagnosed in Patients with Long COVID. Medicina (Kaunas). 2022 Jun 25;58(7):850. doi: 10.3390/medicina58070850. PMID 35888568
- [Background] Umeyama T, Kugimiya T, Ogawa T, Kandori Y, Ishizuka A, Hanaoka K. Changes in cerebral blood flow estimated after stellate ganglion block by single photon emission computed tomography. J Auton Nerv Syst. 1995 Jan 3;50(3):339-46. doi: 10.1016/0165-1838(94)00105-s. PMID 7714328
- [Background] Park HM, Kim TW, Choi HG, Yoon KB, Yoon DM. The change in regional cerebral oxygen saturation after stellate ganglion block. Korean J Pain. 2010 Jun;23(2):142-6. doi: 10.3344/kjp.2010.23.2.142. Epub 2010 May 31. PMID 20556217
- [Background] Kang CK, Oh ST, Chung RK, Lee H, Park CA, Kim YB, Yoo JH, Kim DY, Cho ZH. Effect of stellate ganglion block on the cerebrovascular system: magnetic resonance angiography study. Anesthesiology. 2010 Oct;113(4):936-44. doi: 10.1097/ALN.0b013e3181ec63f5. PMID 20823762
- [Background] Medow MS, Sood S, Messer Z, Dzogbeta S, Terilli C, Stewart JM. Phenylephrine alteration of cerebral blood flow during orthostasis: effect on n-back performance in chronic fatigue syndrome. J Appl Physiol (1985). 2014 Nov 15;117(10):1157-64. doi: 10.1152/japplphysiol.00527.2014. Epub 2014 Oct 2. PMID 25277740
- [Background] Staud R, Boissoneault J, Craggs JG, Lai S, Robinson ME. Task Related Cerebral Blood Flow Changes of Patients with Chronic Fatigue Syndrome: An Arterial Spin Labeling Study. Fatigue. 2018;6(2):63-79. doi: 10.1080/21641846.2018.1453919. Epub 2018 Mar 20. PMID 29707427
- [Background] Jason LA, Gaglio CL, Furst J, Islam M, Sorenson M, Conroy KE, Katz BZ. Cytokine network analysis in a community-based pediatric sample of patients with myalgic encephalomyelitis/chronic fatigue syndrome. Chronic Illn. 2023 Sep;19(3):571-580. doi: 10.1177/17423953221101606. Epub 2022 May 16. PMID 35570777
- [Background] Nkiliza A, Parks M, Cseresznye A, Oberlin S, Evans JE, Darcey T, Aenlle K, Niedospial D, Mullan M, Crawford F, Klimas N, Abdullah L. Sex-specific plasma lipid profiles of ME/CFS patients and their association with pain, fatigue, and cognitive symptoms. J Transl Med. 2021 Aug 28;19(1):370. doi: 10.1186/s12967-021-03035-6. PMID 34454515
- [Background] Giloteaux L, O'Neal A, Castro-Marrero J, Levine SM, Hanson MR. Cytokine profiling of extracellular vesicles isolated from plasma in myalgic encephalomyelitis/chronic fatigue syndrome: a pilot study. J Transl Med. 2020 Oct 12;18(1):387. doi: 10.1186/s12967-020-02560-0. PMID 33046133
- [Background] Wirth K, Scheibenbogen C. A Unifying Hypothesis of the Pathophysiology of Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS): Recognitions from the finding of autoantibodies against ss2-adrenergic receptors. Autoimmun Rev. 2020 Jun;19(6):102527. doi: 10.1016/j.autrev.2020.102527. Epub 2020 Apr 1. PMID 32247028
- [Background] Che X, Brydges CR, Yu Y, Price A, Joshi S, Roy A, Lee B, Barupal DK, Cheng A, Palmer DM, Levine S, Peterson DL, Vernon SD, Bateman L, Hornig M, Montoya JG, Komaroff AL, Fiehn O, Lipkin WI. Metabolomic Evidence for Peroxisomal Dysfunction in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Int J Mol Sci. 2022 Jul 18;23(14):7906. doi: 10.3390/ijms23147906. PMID 35887252
- [Background] Mandarano AH, Maya J, Giloteaux L, Peterson DL, Maynard M, Gottschalk CG, Hanson MR. Myalgic encephalomyelitis/chronic fatigue syndrome patients exhibit altered T cell metabolism and cytokine associations. J Clin Invest. 2020 Mar 2;130(3):1491-1505. doi: 10.1172/JCI132185. PMID 31830003
- [Background] Pongratz G, Straub RH. The sympathetic nervous response in inflammation. Arthritis Res Ther. 2014;16(6):504. doi: 10.1186/s13075-014-0504-2. PMID 25789375
- [Background] Jonsjo MA, Olsson GL, Wicksell RK, Alving K, Holmstrom L, Andreasson A. The role of low-grade inflammation in ME/CFS (Myalgic Encephalomyelitis/Chronic Fatigue Syndrome) - associations with symptoms. Psychoneuroendocrinology. 2020 Mar;113:104578. doi: 10.1016/j.psyneuen.2019.104578. Epub 2019 Dec 26. PMID 31901625
- [Background] Sharma D, Farrar JD. Adrenergic regulation of immune cell function and inflammation. Semin Immunopathol. 2020 Dec;42(6):709-717. doi: 10.1007/s00281-020-00829-6. Epub 2020 Nov 20. PMID 33219396
- [Background] Sugimoto M, Shimaoka M, Taenaka N, Kiyono H, Yoshiya I. Lymphocyte activation is attenuated by stellate ganglion block. Reg Anesth Pain Med. 1999 Jan-Feb;24(1):30-5. doi: 10.1016/s1098-7339(99)90162-1. PMID 9952092
- [Background] Yokoyama M, Nakatsuka H, Itano Y, Hirakawa M. Stellate ganglion block modifies the distribution of lymphocyte subsets and natural-killer cell activity. Anesthesiology. 2000 Jan;92(1):109-15. doi: 10.1097/00000542-200001000-00021. PMID 10638906
- See also: Solve M.E. Ramsay Grant 2022-2023-- Meet the Researchers — https://solvecfs.org/research/ramsay-research-grants/meet-the-researchers/
- See also: Centers for Disease Control and Prevention (CDC). Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Last Reviewed: November 25, 2022 — https://www.cdc.gov/me-cfs/index.html
- See also: ME/CFS clinical trials — https://clinicaltrials.gov/expert-search?term=Myalgic%20Encephalomyelitis%2FChronic%20Fatigue%20Syndrome

DOCUMENTS (1):
  • Informed Consent Form (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05664711/ICF_000.pdf